CLINICAL TRIAL: NCT01151813
Title: Human Behavioral Pharmacology Laboratory (HBPL) Study of Varenicline's Impact on Cocaine and Alcohol Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 811289; K01DA025073 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Dependence; Cocaine Dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): Varenicline, oral administration for 1 week
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Placebo, oral administration for 1 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline, oral target dose of 1.0 mg BID, one week titration.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II within-subjects double-blind placebo-controlled human laboratory study. The purpose of the study is to determine the efficacy of varenicline (Chantix) for reducing cue-induced cocaine and alcohol craving.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and is between 21 and 65 years of age.
2. The subject has used cocaine, alcohol, or cocaine and alcohol at least once per month for at least the past year, and has used cocaine, alcohol, or cocaine and alcohol within the past 30 days.
3. Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
4. Understands and signs the informed consent.

Exclusion Criteria:

1. Meets DSM-IV criteria for current dependence on any substance other than nicotine, cocaine, alcohol or marijuana.
2. Subjects who are currently taking anti-depressant medications (e.g., SSRIs such as citalopram)
3. Patients who are diagnosed during screening with clinical depression using the HAM-D rating scale and present with a score >10.
4. Subjects who are diagnosed with anxiety as diagnosed using the HAM-A anxiety scale with a score >17
5. Subjects who meet current- or lifetime DSM-IV criteria for a psychotic disorder (e.g., schizophrenia)
6. Requires treatment with any psychotropic medication (e.g., antidepressant, antipsychotic, benzodiazepine, or mood stabilizing medication).
7. Subjects who test positive on the urine drug screen for any illicit drugs other than cocaine and marijuana during screening will be allowed a single retest. Those individuals who test positive for amphetamine during screening, given that they provide a copy of a prescription, will only be included if they can safely discontinue amphetamine use for the duration of the study. Subjects will need to provide a urine free of all illicit drugs other than cocaine and marijuana at study onset to be randomized. Subjects who test positive for any drugs other than marijuana prior to a study session will be allowed a single retest and a chance to reschedule their session. If the subject tests positive for any drug other than marijuana at the retest, their participation in the study will be terminated.
8. Use of any investigational medication within the past 30 days.
9. Concomitant use of any one of the following drugs or classes of drugs:

   Anti-depressant drugs such as citalopram, fluoxetine; antipsychotic drugs such as haloperidol; benzodiazepines or other anxiolytic medications; Antihypertensive drugs such as Reserpine, Verapamil; Blood thinners Medications used to treat respiratory diseases such as theophylline; Trimethoprim; Cimetidine; Antiepileptic drugs (AEDs) such as phenytoin or valproic acid.
10. Patients with a known hypersensitivity to varenicline.
11. Patients with severe unstable or serious medical illness such as a seizure disorder, unstable cerebrovascular disease, bronchospastic disease, hyperthyroidism, or diabetes mellitus.
12. Patients with known AIDS or other serious illnesses that may require hospitalization during the study.
13. Female subjects who are pregnant, plan to become pregnant, are currently lactating, or are of child-bearing potential and are not using acceptable methods of birth control; acceptable methods of birth control would include:

    1. Barrier method (diaphragm or condom)
    2. Intrauterine progesterone contraceptive system
    3. Levonorgesterel implant
    4. Medroxyprogesterone acetate contraceptive injection, or
    5. Oral contraceptives.
14. Patients with impaired renal function, as indicated by corrected creatinine clearance below 60 ml/min as determined by the modified Cockcroft equation (CDC, 1986).
15. An unacceptable liver panel (liver function tests; LFTs) that may be indicative of hepatic dysfunction.
16. Clinical laboratory tests (e.g., CBC, blood chemistries, urinalysis) outside normal limits, as determined by PI.
17. History of significant heart disease or dysfunction (e.g., an arrhythmia which required medication, Wolff Parkinson -White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure).
18. Electrocardiography (EKG) indicative of 1st degree heart block, sinus tachycardia, left-axis deviation, non-specific ST or T-wave changes.
19. History of chest pain associated with cocaine use that prompted a visit to a physician.
20. Any medical or psychological condition that could jeopardize the subject's safe participation in the trial as determined by the PI.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline First, Then Placebo: Varenicline, oral target dose of 1.0 mg BID, one week titration; followed by placebo, matched for one week.
- Placebo First, Then Varenicline: Placebo for one week, followed by Varenicline, oral target dose of 1.0 mg BID, one week titration.
Period: Period 1
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Within-subjects Design: Varenicline, oral target dose of 1.0 mg BID, one week titration; placebo, matched for one week. Double-blind counterbalanced order
Arm/Group | Within-subjects Design
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Alcohol Craving
Description: Visual Analog Scale specific to alcohol craving. The VAS has a 100 mm line anchored by 0 and 100. Participants mark the line to indicate how strong their craving is for alcohol. 0 indicates no craving 100 indicates strongest possible craving.
Time Frame: average value over one week
Population: Comparing alcohol craving during Varenicline treatment in participants initially treated with Varenicline (Group 1) to those initially treated with Placebo (Group 2).
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo First, Then Varenicline: Placebo for one week; followed by Varenicline, oral target dose of 1.0 mg BID, one week titration.
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Number analyzed (Participants) | 8 | 7
units on a scale | 20 [0 to 100] | 35 [0 to 100]
Statistical Analysis 1: Comparison: Varenicline First, Then Placebo vs Placebo First, Then Varenicline; Test type: Superiority or Other; p = .02, t-test, 2 sided

2. Primary Outcome: Visual Analog Scale Cocaine Craving
Description: Visual Analog Scale specific to cocaine craving. The VAS has a 100 mm line anchored by 0 and 100. Participants mark the line to indicate how strong their craving is for cocaine. 0 indicated no craving, 100 represents the worst craving imaginable. The subject draws a hatch mark line along the line closer to where there current craving is rated.
Time Frame: average value over one week
Population: Comparing cocaine craving during Varenicline treatment in participants initially treated with Varenicline (Group 1) to those initially treated with Placebo (Group 2).
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Varenicline First, Then Placebo: Varenicline, oral target dose of 1.0 mg BID, one week titration; placebo, matched for one week.
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Number analyzed (Participants) | 8 | 7
units on a scale | 25 [0 to 100] | 65 [0 to 100]
Statistical Analysis 1: Comparison: Varenicline First, Then Placebo vs Placebo First, Then Varenicline; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

3. Primary Outcome: Visual Analog Scale Alcohol Craving 2
Description: Visual Analog Scale specific to alcohol craving. The VAS has a 100 mm line anchored by 0 and 100. Participants mark the line to indicate how strong their craving is for alcohol. 0 indicated no craving, 100 represents the worst craving imaginable. The subject draws a hatch mark line along the line closer to where there current craving is rated. Closer to the 0 means less craving, closer to the 100 means more craving
Time Frame: average over one week
Population: Comparing alcohol craving during Placebo treatment in participants initially treated with Varenicline (Group 1) to those initially treated with Placebo (Group 2).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Number analyzed (Participants) | 8 | 7
units on a scale | 35 [0 to 100] | 55 [0 to 100]
Statistical Analysis 1: Comparison: Varenicline First, Then Placebo vs Placebo First, Then Varenicline; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

4. Primary Outcome: Visual Analog Scale Cocaine Craving 2
Description: Visual Analog Scale specific to cocaine craving. The VAS has a 100 mm line anchored by 0 and 100. Participants mark the line to indicate how strong their craving is for cocaine. 0 indicated no craving, 100 represents the worst craving imaginable. The subject draws a hatch mark line along the line closer to where there current craving is rated. Closer to the 0 means less craving, closer to the 100 means more craving
Time Frame: average over one week
Population: Comparing cocaine craving during Placebo treatment in participants initially treated with Varenicline (Group 1) to those initially treated with Placebo (Group 2).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Varenicline First, Then Placebo | Placebo First, Then Varenicline
Number analyzed (Participants) | 8 | 7
units on a scale | 65 [0 to 100] | 80 [0 to 100]
Statistical Analysis 1: Comparison: Varenicline First, Then Placebo vs Placebo First, Then Varenicline; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: through study completion, two weeks
Description: Participants were asked to report adverse events at each study visit by nurses using a checklist of known (previously reported) adverse events, as well as novel adverse events.
Groups:
- Varenicline: While receiving Varenicline, oral target dose of 1.0 mg BID, one week titration
- Placebo: While receiving Placebo, one week
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=15) | Placebo (N=15)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No